CLINICAL TRIAL: NCT00387153
Title: Phase 1 OL, Dose Escalating, Multiple Dose Study To Determine The Safety, Tolerability, MTD, And Pharmacokinetics Of MPC-2130 Administered As Daily IV Infusions For 5 Days, Repeated Every 21 Days, In Patients With Refractory Cancer
Brief Title: Phase 1 Clinical Trial MPC-2130 Treatment of Blood Cancers / Refractory Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Last subject enrolled experienced bradycardia; study was terminated by Sponsor.
Sponsor: Myriad Therapeutics, Inc. (Industry)
Responsible Party: Richard Wenstrup, Myriad Therapeutics, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPC-2130-04-002
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Results first posted 2009-10-22 (Estimated); Last update posted 2009-11-03 (Estimated); Status verified 2009-10

CONDITIONS: Cancer
Keywords: Oncology; Cancer; Blood Cancers
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: MPC-2130 — MPC-2130 10 mg/mL administered by intravenous infusion over 1-2 hours

SUMMARY:
Phase 1 Open-label treatment with MPC-2130 for subjects with refractory cancer.

DETAILED DESCRIPTION:
MPC-2130 Phase 1 Clinical study was designed to evaluate its safety and pharmacokinetic profile in patients with advanced metastatic tumors or blood cancers as well as refractory cancers that progressed despite previous chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Be capable of understanding the informed consent form (ICF) and complying with the protocol, and must sign the ICF prior to the performance of any study related procedures;
2. Have cancer that is nonresponsive despite prior treatment with current standard of care regimens or for whom there are no available effective therapies;
3. Have measurable or evaluable neoplastic disease;
4. Be greater than or equal to age 18;
5. Have and ECOG Performance Status score of less than or equal to 2;
6. Have adequate organ function defined by:

   1. Liver function tests (AST & ALT) less than or equal to 3 times the upper limit of normal (ULN);
   2. Bilirubin less than or equal to 1.5 X ULN;
   3. Serum Creatinine less than or equal to 1.5 X ULN;
   4. Hemoglobin greater than or equal to 8.0 g/dL;
7. Have recovered or stabilized from clinically significant toxicities of prior chemotherapy, surgery, or radiotherapy;
8. Have left ventricular ejection fraction (LVEF) of greater than or equal to 45% by multiple gated acquisition (MUGA) scan or echocardiogram.

Exclusion Criteria:

1. Have had a prior serious, uncontrollable hypersensitivity reaction to Cremophor EL;
2. Be pregnant or lactating (women of childbearing potential must use appropriate birth control (abstinence, barrier methods, oral contraceptives and/or intrauterine devices) during the entire duration of the study, or the patient must be surgically sterile (with documentation in the patient's medical records);
3. Receive any other anticancer treatment or investigational therapy within 14 days prior to day 1; or within 6 weeks after prior mitomycin C or nitrosourea. Patients with advanced prostate cancer may continue to receive leutinizing hormone-releasing hormone (LHRH) therapy while in this study;
4. Have previously enrolled in this trial. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-08; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Wenstrup, MD, Study Director — Myriad Therapeutics, Inc.
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- MPC-2130 Group 1: Group 1 will be dosed at 10 mg/ml administered via IV over a 1-2 hour period.
Period: Overall Study
Arm/Group | MPC-2130 Group 1
Started | 8
Completed | 0
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Disease Progression | 3
Not completed — Lack of Response | 4

BASELINE CHARACTERISTICS:
Arm/Group | MPC-2130 Group 1
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 48.5 (21.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Dose Limiting Toxicities and Grade 3/4 Adverse Events. As a General Guideline, a Severe Adverse Event is Considered Grade 3, and a Life Threatening or Disabling Adverse Event is Considered Grade 4.
Description: Dose limiting toxicities include any grade 3 nonhematological toxicity(excluding nausea/vomiting or alopecia); greater than grade 3 nausea/vomiting uncontrolled by aggressive antiemetic support; grade 4 neutropenia lasting more than 5 days, or any febrile (38.5° C or 101° F) grade 3/4 neutropenia; grade 4 thrombocytopenia.
  An adverse event is any reaction, side effect, or other untoward event, regardless of relationship to MPC-2130 that occurs any time after the beginning of the first IV infusion of MPC-2130 until 30 days after MPC-2130 discontinuation.
Time Frame: First 21 days on treatment (Cycle 1)
Population: A total of 8 subjects were enrolled in the study. Statistical analyses were intended to be descriptive since the goal for the study was to determine the maximum tolerated dose and general safety and tolerability of MPC-2130.
Measure: Number; unit: Participants
Arm/Group | MPC-2130 Group 1
Number analyzed (Participants) | 8
Participants | 8

2. Primary Outcome: Pharmacokinetics
Description: Characterization of MPC-2130 pharmamcokinetics consisting of AUC, tmax, Cmax, half-life and clearance.
Time Frame: First 5 days of treatment (Cycle 1)
Reporting Status: Not Posted

3. Secondary Outcome: Antiproliferative Activity
Description: Observation for any evidence of antiproliferative activity of MPC-2130 in treatment of a variety ofrefractory neoplasias.
Time Frame: Every 42 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | MPC-2130 Group 1
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MPC-2130 Group 1 (N=8)
sinus bradycardia (Cardiac disorders) | 1 (1)
disease progression (Blood and lymphatic system disorders) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MPC-2130 Group 1 (N=8)
blood and lymphatic system disorders (Blood and lymphatic system disorders) | 5 (6)
Cardiac disorders (Cardiac disorders) | 2 (2)
gastroinstestinal disorders (Gastrointestinal disorders) | 7 (17)
general disorders and administration site conditions (General disorders) | 6 (16)
hepatobiliary disorders (Hepatobiliary disorders) | 1 (1)
immune system disorders (Immune system disorders) | 1 (1)
infection and infestations (Infections and infestations) | 4 (7)
contusion (Injury, poisoning and procedural complications) | 1 (1)
investigations (Investigations) | 7 (8)
metabolism and nutrition disorders (Metabolism and nutrition disorders) | 8 (23)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
nervous system disorders (Nervous system disorders) | 7 (16)
psychiatric disorders (Psychiatric disorders) | 5 (9)
respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3 (7)
skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 5 (6)
vascular disorders (Vascular disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right to the 1st publication within 12 months of study conclusion. After, the institution/PI may publish data after submission to the sponsor for review.